CLINICAL TRIAL: NCT04532944
Title: Exploring in Vivo the Energetic Origin of Neurodegeneration in Multiple Sclerosis: a Ultra-high Field Sodium Imaging, Phosphorus Spectroscopy and Diffusion-weighted Spectroscopy Study.
Brief Title: The Energetic Origin of Neurodegeneration in MS
Acronym: ENERGYSEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C19-20; 2019-A01931-56 (Registry Identifier: ID RCB)
Record Dates: First submitted 2020-07-30; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: energy dysfunction; neurodegeneration; 7 T MRI; sodium imaging; phosphorus spectroscopy; diffusion-weighted spectroscopy
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: 40 patients with MS and 15 healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with MS (Other): 20 relapsing-remitting and 20 progressive MS patients
  Interventions: Diagnostic Test: imaging of energy dysfunction
- healthy controls (Other): 15 age- and sex-matched healthy controls
  Interventions: Diagnostic Test: imaging of energy dysfunction

INTERVENTIONS:
Diagnostic Test: imaging of energy dysfunction — 7T sodium imaging, phosphorus spectroscopy and 3T diffusion-weighted spectroscopy

SUMMARY:
In multiple sclerosis (MS), the sequence of events leading to irreversible neuro-axonal degeneration, which is a major determinant of clinical disability, is poorly understood. Recently, the key role of neuronal energy dysfunction in driving axonal degeneration has been highlighted. In the neuronal injury pathway triggered by inflammation and myelin disruption, multiple adaptive changes force the neuron to a temporary condition of "virtual hypoxia", characterized by a mismatch between energy demand and supply. If this condition of energy dysregulation is not reversed within an appropriate time-window, neurons enter an irreversible axonal degeneration.

Two key questions on the relationship between early energy dysregulation and neurodegeneration remain unanswered:

i) whether brain energy dysfunction measured at a given time point can predict the subsequent occurrence of neurodegeneration; ii) to what extent and for how long neurons can bear this "virtual hypoxia" before undergoing structural damage.

Tracking the "energetic signature" of MS and defining its temporal distance from irreversible damage is essential for the development of neuroprotective therapies.The recent optimization of innovative magnetic resonance (MR)-based techniques such as sodium (23Na) MRI, phosphorus MR spectroscopy (31P-MRS), and diffusion-weighted 1H MRS (DW-MRS) has allowed the generation of promising in vivo data on cellular energy dysregulation in MS.

The main objective of this project is to explore whether MR-derived metrics of energy dysregulation predict MR-derived parameters of cortical neurodegeneration developing over 2 years, as reflected by cortical atrophy. To address this key question, the Investigators will use a combination of 23Na MRI, 31P MRS, and DW-MRS associated with advanced MRI sequences to explore energy dysregulation in the sensorimotor region, and measurements of cortical atrophy in the same area after 24 months in 40 patients with either relapsing-remitting or progressive MS and 15 age- and gender-matched healthy controls.

The Investigators will also test whether MR-derived metrics of energy dysregulation at study entry correlate, both cross-sectionally and longitudinally, with: i) global cortical atrophy; ii) functional cortical reorganization resulting from the condition of energy dysregulation, which precedes the occurrence of structural damage; iii) cortical demyelination and remyelination; iv) clinical, neuropsychological and biological measures.

DETAILED DESCRIPTION:
1. RESEARCH JUSTIFICATION

1.1 Energy dysregulation is a key process in the physiopathology of neurodegeneration in MS

Several mechanisms have been suggested to play a major role in the physiopathology of neurodegeneration in multiple sclerosis (MS), among which: inflammatory demyelination, excitotoxicity, oxidative stress and ionic channel dysfunction. Each of these mechanisms is potentially implicated in inducing an energy dysregulation. Moreover, the notion that early neuronal energy failure may play a key role in axonal degeneration is being more and more acknowledged. In these physiological conditions, myelin sheath integrity not only allows efficient saltatory conduction of the action potential, but it also helps to maintain the environment for neuronal survival by assuring the correct amount of cellular energy.

Following myelin disruption and inflammation, multiple adaptive changes force the neurone to enter a temporary state of "virtual hypoxia". Indeed, the loss of axonal coverage determines the VGSC redistribution along the axon and the re-expression of NaV1.2.

Furthermore, demyelination induces mitochondrial proliferation along damaged axons, together with a complex for hyperactivity in order to support the sodium/potassium pump. These compensatory mechanisms initially overcome the conduction block resulting from demyelination, but in such conditions transmembrane electrochemical gradients are maintained at the cost of an increased energy demand.

This supplementary energy demand leads to a dysequilibrium between energy demand and supply, called "neuronal virtual hypoxia". In MS energetic distress is worsened by the inflammatory environment, which affects mitochondrial function and is associated with a cell structural deformation. This condition of energy dysfunction is potentially reversible in the first stages of the disease but, if not reversed after a certain time it induces a cascade characterised by a mitochondrial function failure, free radical production and sodium/potassium ATPase dysfunction. Ionic pump dysfunction induces an accumulation of inter-cellular sodium with an inversion of calcium flux operated by the Na+/Ca2+ pump. Calcium intracellular influx eventually leads to an irreversible neuronal degeneration. Therefore, identifying in-vivo the early phase of neuronal energy dysfunction proceeding neuro-axonal death and understanding its temporal relationship with reversible neuronal degeneration is essential for the development of therapies aimed at reverting this degenerative process and maintain long term neuronal integrity.

1.2 Imaging energy dysregulation: state of the art

The optimisation over the past few years of innovative techniques based on magnetic resonance (MR) such as sodium MRI (23Na), phosphorus spectroscopy (31P-MRI) and diffusion-weighted spectroscopy (DW-MRS), have enabled the production of promising data which allow the clarification of different aspects of the initial phase of energy dysregulation in MS.

Several studies using 23Na MRI have shown an increase of the concentration of total sodium in the brain of patients with MS, which is correlating with clinical disability. More recently, more sophisticated techniques to quantify 23Na concentration have been proposed, such as "triple quantum filtered (TQF) imaging", which allows the differentiation between intracellular and extracellular sodium, thus providing unique information on the early phase of energy dysregulation. Due the relatively weak sensibility of 23Na MRI, high-field MRI is particularly suited for TQF. The team lead by professor Matilde Inglese has recently applied 7 tesla TQF imaging in MS, showing that patients with a relapsing/remitting form of the disease (RR-MS) have increased intracellular sodium concentration compared to healthy volunteers. This reflects the pathological intracellular accumulation of 23Na as a consequence of Na+ K+ ATpase dysfunction.

31-MRS allows the direct measurement of the concentration in the brain of phosphocreatine (PCr) and adenosine triphosphate (ATP), which is the main energy currency of cells. 31P-MRS at 3T has shown that MS patients present higher PCr levels in the normal-appearing white matter when compared to healthy controls. 21P-MRS has also shown that beta-ATP percentage was higher in RR-MS and lower in progressive forms, reflecting a "relatively high energy state" in the early phases of the disease, with a reduction in the progressive phase, leaving room for axonal degeneration.

Important technical processes have been reached through the successful generation of 31P-MRS data at 7T.

DW-MRS gives in-vivo measurements of the diffusion properties of creatine (Cr) + PCr. In a recent study using DW-MRS at 3T, the Investigators found a reduced Cr+PCr diffusivity in the normal-appearing white matter and the thalami of patients with MS compared with healthy controls, reflecting a reduction of energy reserved in neurons and glial cells. Two alternative hypotheses could explain the observed reduction of Cr+PCr diffusivity: an altered intracellular transport of creatine, in particular from oligodendrocytes to neurones from one to another, or a reduced PCr consumption due to an altered function of creatine kinase B.

Overall, these results confirm the strong potential of combining these different techniques (23Na MRI, 31PMRS and DW-MRS) in order to obtain innovative information on each aspect of the pathogenic cascade linking energy dysregulation to neuro-axonal degeneration in MS.

2. OBJECTIVES

2.1 Main objective

The main objective of this project is to explore the relationship between the MRI-derived parameters reflecting energy dysregulation in the motor sensory regions (MSR) at study entry, and the parameters of neurodegeneration in the MSR after 24 months in RR-MS and PMS patients compared to healthy volunteers, through a combination of 23Na quantitative MRI, 31P-MRS and DW-MRS, and measurements of cortical thickness.

2.2 Secondary objectives

The secondary objectives of this research will be:

(i) To compare MRI-derived metrics of energy dysregulation between patients and controls in the whole brain and the MSR at study entry.

(ii) To define the correlations between MRI-derived metrics of energy dysregulation and cortical demyelination at study entry, as well as cortical myelination after 12 months.

(iii) To study the correlation between cortical 23Na MRI at study entry and the evolution of cortical volume over 24 months.

(iv) To study the correlations between MRI-derived metrics of energy dysregulation and early axonal damage a well as axonal-dendritic density in the whole brain and in the MSR: 1) at study entry; 2) over the follow-up period of 24 months.

(v) To study the relationship between MRI-derived metrics of energy dysregulation and the changes of brain connectivity at study entry, at 12 and 24 months.

(vi) To establish the correlations between MRI-derived metrics and serum neurofilaments measured at study entry, at 12 and 24 months.

(vii) To establish the contribution of MRI-derived metrics of energy dysregulations to clinical disability and to cognitive dysfunction, at study entry and at 24 months.

3. CONCEPTION OF THE RESEARCH PROJECT

3.1 Type of research project

This is a monocentric research project on human beings with physiopathologic purposes (no health products involved), with a duration of 24 months, whose aim is to explore the role of energy dysregulation in neurodegeneration, which is the main pathologic substrate of clinical progression in patients with MS. Our aim is to investigate the relationship between energy dysfunction and neuro-axonal damage in patients with MS compared to healthy controls, using a combination of imaging methods and clinical, cognitive and biological tests.

Given that the techniques used in the study involve imaging methods with the injection of contrast agents, the research will be classified as interventional research of category 1, according to the Jardé Law.

3.2 Methodology of the research

This is a non-randomized, controlled, open label clinical-radiological research.

Patients will be selected from the cohorts followed at the Department of Neurology of Saint-Antoine Hospital and the Department of Nervous System Pathologies of the Pitié-Salpêtrière Hospital. They will receive a first information on the research during the consultation, and the information form may be delivered on this occasion.

Healthy volunteers will be selected from the volunteers of the Center of Clinical Investigation (CIC) of the Pitié-Salpêtrière Hospital.

All participants will be included at the CIC of the Brain and Spine Institute (ICM) - Pitié-Salpêtrière Hospital.

A group of RR-MS (n=20) and progressive (PP-MS or SP-MS, n=20) patients will be studied and compared to a group of healthy volunteers (n=15), age- and gender-matched (but without a 1:1 matching between patients and controls). The choice of matching a sample of 40 patients to a sample of 15 healthy volunteers is based on the calculation of the minimum number of observations per group needed to detect a between-group difference in the evaluation criteria, using a multivariable linear regression model.

Each patient and healthy volunteer will undergo four visits:

Visit 1 (inclusion visit) - D0 : ICM (CIC/CENIR) (30-minute clinical visit + 65-minute 3 T MRI)

* information, verification of inclusion/exclusion criteria, signature of the informed consent form
* neurological evaluation (EDSS, MRC scores) and testing of fatigue (MFIS, Jamar hydraulic hand dynamometer) to assess the level of physical impairment
* neuropsychological tests (BICAMS) to evaluate the level of cognitive impairment
* pregnancy test for all women of child-bearing age
* 3T MRI - with gadolinium injection for patients only (see 8.1 for administration procedures) - with DW-MRS sequences to quantify tCr et NAA (N-acetyl aspartate) diffusivity in a voxel centered on the MSR, and with sequences for volumetric, structural and functional analyses (65 min)
* blood sampling (4 mL) to search for neurofilaments as biological markers of neurodegeneration.

Visit 2 - M1: NeuroSpin (CEA Center in Saclay, Gif-sur-Yvette, France) (120 minutes)

* Urinary pregnancy test for all women of child-bearing age
* 7T MRI including a whole brain 23Na MRI and a 31P MRS centered on the MSR voxel for sodium, ATP and PCr quantification (1h40min)

Visit 3 - M12 : ICM (CIC/CENIR) (15-minute clinical visit + 65-minute 3 T MRI)

* neurological evaluation (EDSS, MRC scores) and testing of fatigue (MFIS, Jamar hydraulic hand dynamometer) to assess the level of physical impairment
* pregnancy test for all women of child-bearing age
* 3T MRI - using the same protocol of V1 - with gadolinium injection for patients only (see 8.1 for administration procedures) - with DW-MRS sequences to quantify tCr et NAA (N-acetyl aspartate) diffusivity in a voxel centered on the MSR, and with sequences for volumetric, structural and functional analyses (65 min)
* blood sampling (4 mL) to search for neurofilaments as biological markers of neurodegeneration.

Visit 4 - M24 : ICM (CIC/CENIR) (30-minute clinical visit + 65 minute 3 T MRI)

* neurological evaluation (EDSS, MRC scores) and testing of fatigue (MFIS, Jamar hydraulic hand dynamometer) to assess the level of physical impairment
* neuropsychological tests (BICAMS) to evaluate the level of cognitive impairment
* pregnancy test for all women of child-bearing age
* 3T MRI - using the same protocol of V1 - with gadolinium injection for patients only (see 8.1 for administration procedures) - with DW-MRS sequences to quantify tCr et NAA (N-acetyl aspartate) diffusivity in a voxel centered on the MSR, and with sequences for volumetric, structural and functional analyses (65 min)
* blood sampling (4 mL) to search for neurofilaments as biological markers of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria for MS:

1. RR-MS patients with a disease duration of less than 10 years:

   * 18-55 years
   * clinically defined RR-MS according to the 2017 revised McDonald's criteria (MS diagnostic criteria 2017)
   * disease duration <10 years
   * ability to understand the research objectives and the procedure details, and to sign the informed consent
   * affiliation with the French National Health Insurance, Universal Medical Coverage (CMU) or any equivalent
2. Patients with progressive MS (primary or secondary) of less than 10 years:

   * 18-55 years
   * clinically defined progressive MS according to the 2017 revised McDonald's criteria
   * disease duration <10 years from the beginning of the progressive phase
   * ability to understand the research objectives and the procedure details, and to sign the informed consent
   * affiliation with the French National Health Insurance, Universal Medical Coverage (CMU) or any equivalent

Inclusion Criteria for healthy controls:

* 18-55 years (matched with patients)
* no known general pathologies
* ability to understand the research objectives and the procedure details, and to sign the informed consent
* affiliation with the French National Health Insurance, Universal Medical Coverage (CMU) or any equivalent

Exclusion Criteria for MS:

* Pregnant or breastfeeding women
* Last infusion of cyclophosphamide, mitoxantrone or methylprednisolone realized less than 1 month before inclusion
* last clinical relapse less than one month before inclusion
* severe cardiac, pulmonary, hepatic, hematologic renal, gastrointestinal disease, or cancer
* contraindications to MRI: claustrophobia, pace-maker implant, any surgical ferromagnetic clips, ocular implants, any intraocular or intracranial metallic fragments, any metallic objects able to concentrate the radiofrequency field, cochlear implants, cardiac or brain stimulators, any tattoos or permanent makeup on the face, renal failure (exclusion criterion for gadolinium injection) patients not willing to be informed of any possible cerebral malformations incidentally discovered at the MRI exam
* severe renal failure (clearance of creatinine < 30ml/min)
* history of allergic reactions to gadolinium salts
* any other chronic neurological disorders associated
* persons deprived of liberty by law or by administrative decision
* Persons under legal protection

Exclusion Criteria for healthy controls:

* Pregnant or breastfeeding women
* severe cardiac, pulmonary, hepatic, hematologic renal, gastrointestinal disease, or cancer
* contraindications to MRI : claustrophobia, pace-maker implant, any surgical magnetic clips, ocular implants, any intraocular or intracranial metallic fragments, any metallic objects able to concentrate the radiofrequency field, cochlear implants, cardiac or brain stimulators, any tattoos or permanent makeup on the face
* person not willing to be informed of any possible cerebral malformations incidentally discovered at the MRI exam
* associated chronic neurological disorders
* persons deprived of liberty by law or by administrative decision
* Persons under legal protection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Energy dysregulation in the whole brain with sodium imaging | 0-12 months
  Evaluation of the levels of total, intracellular and extracellular sodium quantified through 23Na MRI in the whole brain.
Energy dysregulation in the motor-sensory region (MSR) with phosphorus spectroscopy | 0-12 months
  Evaluation of ATP and PCr concentrations measured through 31P MRS in a voxel centred on the left MSR
Energy dysregulation in the motor-sensory region with diffusion-weighted spectroscopy | 0-12 months
  Evaluation of the ADC of tCr (Cr + PCr) measured through DW-MRS in a voxel centred on the left MSR.
Neurodegeneration in the MSR after 24 months | 0-24 months
  Neurodegeneration after 24 months will be evaluated by the measurements of the following parameters:
  Evaluation of MSR cortical thickness after 24 months and relative change in MSR cortical thickness between study entry and 24 months measured with Freesurfer (https://surfer.nmr.mgh.harvard.edu).

SECONDARY OUTCOMES:
Patient-specific profiles of energy dysregulation | 0-12 months
  The difference of MRI-derived metrics of energy dysregulation between patients and controls at study entry will be evaluated with 23Na MRI in the whole brain, and with 23Na MRI, 31P MRS and DW-MRS in the MSR
cortical demyelination and remyelination | 0-12 months
  Cortical demyelination at study entry will be measured by cross-sectional cortical magnetisation transfer ratio (MTR), and cortical remyelination after 12 months will be evaluated by the measurement of cortical MTR change over 12 months
neuro-axonal damage over time | 0-12-24 months
  Early axonal damage will be quantified through the NODDI-derived metrics
functional changes in brain connectivity | 0-12-24 months
  Changes in brain connectivity at study entry and after 12 and 24 months will be measured by resting-state functional MRI
serum markers of tissue damage | 0-12-24 months
  Serum neurofilaments, measured at study entry and at 12 and 24 months, will be used as a biomarker of acute and chronic neuronal lesions
physical and cognitive dysfunction | 0-12-24 months
  Neurologic disability will be evaluated by EDSS
physical and cognitive dysfunction | 0-12-24 months
  Neurologic disability will be evaluated by MFIS
physical and cognitive dysfunction | 0-12-24 months
  Neurologic disability will be evaluated by BICAMS

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04532944/Prot_SAP_000.pdf